CLINICAL TRIAL: NCT05731531
Title: Gastric Myoelectric Activity With Water Load Satiety Test as a Predictor of Individual Successful Response to Treatment by Various Bariatric Procedures.
Brief Title: EGG Test as a Predictor for an Individual Response to Treatment by Various Bariatric Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rakesh Kalapala, Director Endoscopy (center for obesity and metabolic therapy), Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AIG/IEC-BH&R32/07.2022-02
Record Dates: First submitted 2022-11-14; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Bariatric Surgery; Gastric Motor Dysfunction; Gastroparesis
Keywords: Bariatric surgery; Electrogastrography; Gastric Myoelectric activity
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- Group A (Other): Group of 50 patients who undergo BIG placement
  Interventions: Device: ELECTROGASTROGRAPHY
- Group B (Other): Group of 50 patients who undergo endoscopic sleeve gastroplasty
  Interventions: Device: ELECTROGASTROGRAPHY
- Group C (Other): Group of 50 patients who undergo Surgical sleeve gastrectomy
  Interventions: Device: ELECTROGASTROGRAPHY
- Group D (Other): Group of 50 patients who undergo RYGB
  Interventions: Device: ELECTROGASTROGRAPHY
- Group E (Other): Group of 50 healthy subjects
  Interventions: Device: ELECTROGASTROGRAPHY

INTERVENTIONS:
Device: ELECTROGASTROGRAPHY — Electrogastrography as a new tool to customize choice of Bariatric therapies by determining success or failure based on GMA and WLST results has not been studied. GMA measures the normal or depleted gastric ICCs and the WLST measures gastric capacity, objective measures that may be important to predict success of Bariatric procedures and thus to help with patient selection to maximize efficacy and minimize side effects.

SUMMARY:
Total body weight loss (TBWL) after bariatric endoscopy (BE) is variable. Gastric emptying may be normal, rapid or delayed in patients with obesity and be a factor in variable BE outcomes. Gastric myoelectrical activity (GMA) reflects gastric pacemaker activity which controls gastric contractions. The non-invasive electrogastrogram(EGG) uses standard electrodes positioned on the abdominal surface to record GMA. The investigators postulate that GMA patterns recorded with EGG will reflect subgroups in regards to stomach electrical physiology in obesity and that these subgroups will be useful in selecting patients for various BE procedures to maximize success of the procedures.

DETAILED DESCRIPTION:
Electrogastrography is a non-invasive method of recording GMA that is used to diagnose gastric dysrythmias in patients with intractable chronic nausea and vomiting, gastroparesis and gastroesophageal reflux.

Bariatric Techniques: 3 categories 1)restrictive,2) mal absorptive 3)mixed Bariatric endoscopy techniques have emerged as safe and effective treatment that include restrictive endoscopic techniques: Intragastric balloons or endoscopic sleeve gastroplasty(ESG),primary surgery obesity endoluminal (POSE) or Endo-sleeve (GESP or POSE 2.0) procedures; malabsorptive techniques :endoluminal bypass (endobarrier),duodenal mucosa resurfacing; extraction methods (Aspire); electrical stimulation : gastric pacemaker, vagal blockage and other procedures.

Weight loss and long-term maintenance may be conditioned by changes in GMA, as well as by anatomical modifications induced by the bariatric procedure.

Since anatomical modifications of the stomach by the BE procedures are related to weight loss, The purpose is to determine whether different procedures to reduce gastric capacity will result in substantial changes in GMA and in the water load volume ingested. No studies that have studied obese population before and after such BE procedures are available.

Therefore, whether obese patients have the GMA that is similar to those with functional dyspepsia and normal weight . Also, the usefulness of electrogastrography as a new tool to customize choice of Bariatric therapies by determining success or failure based on GMA and WLST results has not been studied. GMA measures the normal or depleted gastric ICCs and the WLST measures gastric capacity, objective measures that may be important to predict success of Bariatric procedures and thus to help with patient selection to maximize efficacy and minimize side effects.

Demonstrate the usefulness of EGG meizuring the GMA by identifying subtypes with the Water Load Satiety Test (WLST) in obese adults to predict individual successful responses to BE treatments: Intragastric Balloon (IGB) placement and Apollo Endoscopic Sleeve Gastroplasty (ESG) method

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged between 18-65 yrs
* IMC basal ≥ 30 kg/m2
* Patient undergoing bariatric intervention willing to participate in the study
* Informed consent (oral and written) for the tests to be carried out.

Exclusion Criteria:

* Presence of severe cardiac, renal, hepatic, or neurological disease
* Long term use of medication that alter gastric motility (> 4 weeks)
* Significant alcohol or opioids or narcotics or tobacco
* Active malignancy 5.Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in EGG parameters like WLST (water load satiety test) GMA Gastric myoelectric activity),Predominant frequency of stomach. | 1st or 3rd month of baritaric surgery
  Pre-intervention EGG parameters and/or changes in EGG parameters (one/three months) after bariatric intervention can predict clinical success at the end the of follow up
Changes in EGG parameters like WLST (water load satiety test) GMA Gastric myoelectric activity),Predominant frequency of stomach at end of the follow up. | 18-24 month
  Pre-intervention EGG parameters and/or changes in EGG parameters (one/three months) after bariatric intervention can predict clinical success at the end the of follow up

SECONDARY OUTCOMES:
EGG as a diagnostic tool to measure WLST (water load satiety test) GMA Gastric myoelectric activity),Predominant frequency of stomach. | 12-18 months
  EGG is a feasible diagnostic tool in obese population with reproducible and predictible results

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Kalpala, MBBS,MD,DM, Study Director — Senior consultant
Locations (1):
- AIG Hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kral J, Machytka E, Horka V, Selucka J, Dolecek F, Spicak J, Kovarova V, Haluzik M, Buzga M. Endoscopic Treatment of Obesity and Nutritional Aspects of Bariatric Endoscopy. Nutrients. 2021 Nov 26;13(12):4268. doi: 10.3390/nu13124268. PMID 34959819
- [Background] Jirapinyo P, Thompson CC. Endoscopic Bariatric and Metabolic Therapies: Surgical Analogues and Mechanisms of Action. Clin Gastroenterol Hepatol. 2017 May;15(5):619-630. doi: 10.1016/j.cgh.2016.10.021. Epub 2016 Oct 28. PMID 27989851

DOCUMENTS (1):
  • Study Protocol (2022-07-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT05731531/Prot_000.pdf